CLINICAL TRIAL: NCT06569641
Title: Cardiac Surgery Recovery in Infants Assessed Using Neoneur Feeding System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neoneur LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C03101
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Disease; Post-Surgical Complication; Cardiac Disease
Keywords: Recovery
MeSH Terms: conditions — Infant, Newborn, Diseases; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Infant feeding patterns during standard care. The Neoneur Feeding System captures data such the changes in these feeding patterns can be measured. This study is capturing longitudinal changes over a short period of time, to see if they reflect infant recovery from surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Feeding Assessment (Experimental): While Feeding, use Neoneur Feeding System to measure feeding patterns (suck, swallow, and breathing)
  Interventions: Device: Neoneur Feeding System

INTERVENTIONS:
Device: Neoneur Feeding System — The Neoneur Feeding System is placed between a nipple and a bottle, and used to measure feeding skill patterns.

SUMMARY:
A prospective non-randomized longitudinal design of 30-40 infants from initiation of oral feeding until discharge to track feeding changes as a potential indicator of surgical recovery.

DETAILED DESCRIPTION:
Safe oral feeding is a challenge for infants born with complex congenital heart disease (CHD). These infants are likely to require tube-assisted feeding at the initiation of enteral feeding and struggle to transition to full oral feeding. Infant post-surgery recovery includes a safe transition to oral feeding without respiratory risk. Neoneur Feeding System, consists of a novel hand-held, mobile phone application, and a cloud based computation, which innovatively measures patterns of oral cavity pressure synchronized with respiration, providing a quantitative assessment of feeding patterns. Yet there has been no quantitative means of measuring this recovery process. The concept of post-surgical recovery model is not new. The adult literature is replete with physiologic and behavioral indicators of recovery. More recently Roy and colleagues introduced a recovery model for post-surgical CHD children to adults using a component metrics of physiologic parameters. We are proposing to develop an infant specific recovery model using feeding patterns using data generated by the Neoneur device. The model, using the lens of behavioral organization, will include feeding measurements from initiation of oral feeding to discharge.

This study will evaluate the association between feeding recovery and clinical assessment of infant behaviors as measured in a brief survey to assess irritability, ability to be soothed, alertness, non-nutritive sucking, and muscle tone. Forty infants will be recruited from the PCICU-CSD at MUSC to capture thirty usable infant sets of Neoneur data from the PCICU-CSD at MUSC. This data will be assessed using the Neoneur Feeding System to create a model of feeding recovery.

ELIGIBILITY:
Inclusion Criteria:

* Complex congenital heart disease requiring cardiac surgery during first month of life
* Gestational age>=35 weeks at birth

Exclusion Criteria:

* No other major non-cardiac congenital anomalies,
* No history of major neurologic insult
* Not listed for a heart transplant,
* Not intubated for >4 weeks post-surgery,
* Not trisomy 13, 18, and 21
* No cleft lip/palate.

Ages: 1 Day to 50 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
To test the validity in use of feeding parameters to measure recovery progress for infants with complex CHD | 12 months
  A comparison of feeding patterns (oral cavity pressure changes in suck and swallow, and respiratory patterns) and changes as an infant recovers and determination if there is a greater than 60% concordance with behavioral survey measuring recovery.

SECONDARY OUTCOMES:
Comparison of Neoneur Feeding system measurements seen in post surgical infants, to match clinical observation of suck, swallow, and breathing during oral feeding. | 12 months
  70% concordance between Neoneur Feeding Trace, and clinical observation

IPD SHARING:
Plan to Share IPD: No
All Protocol, Inform Consent, and Final data will be shared with the research sites for their use in publications, and as required by the NIH.